CLINICAL TRIAL: NCT00403364
Title: Sequential Therapy Versus Triple Therapy for Helicobacter Pylori Eradication: a Placebo-controlled Trial
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1112/2006; No grant received
Record Dates: First submitted 2006-11-22; First posted 2006-11-23 (Estimated); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori infection; Treatment; Double blind placebo controlled trial

INTERVENTIONS:
Drug: Placebo amoxicillin pantoprazole clarithromycin tinidazole

SUMMARY:
To assess if a sequential treatment regimen better eradicates H. pylori than does a triple drug regimen in adults with dyspepsia or peptic ulcer disease.

DETAILED DESCRIPTION:
Background: Antimicrobial resistance has decreased eradication rates for H. pylori worldwide.

Objective: To assess if a sequential treatment regimen better eradicates H. pylori than does a triple drug regimen in adults with dyspepsia or peptic ulcer disease.

Design: Placebo-controlled trial. Setting: Two Italian Hospitals between September 2003 and April 2006. Patients: 300 dyspeptic or peptic ulcer patients Measurements: 13C urea breath test, upper endoscopy, histology, rapid urease test, bacterial culture, and antibiotic resistance assessment.

Intervention: 10-day sequential regimen (pantoprazole 40 mg, amoxicillin 1 g plus placebo for the first 5 days, followed by pantoprazole 40 mg, clarithromycin 500 mg and tinidazole 500 mg for the remaining 5 days) in 150 patients or standard 10-day therapy (pantoprazole 40 mg, clarithromycin 500 mg, and amoxicillin 1 g) in 150 patients. All drugs were given twice daily.

Results: There were 295 patients (Intent to treat) of whom 91% (95% CI: 86.5-95.7) had successful eradication with sequential therapy compared to 78% (95% CI: 71.2-84.5) for standard therapy (difference: 13.3%; 95%). The sequential therapy was significantly more effective in patients with clarithromycin resistant strains (88.9% patients vs. 28.6%; P = 0.0034). The incidence of major and minor side effects did not differ between therapy groups (17% vs. 17%).

Limitations: Follow-up was incomplete in 4.6% and 2.7% patients in sequential and standard therapy, respectively. The higher efficacy of sequential regimen should be confirmed outside Italy.

Conclusions: Sequential therapy is superior to conventional therapy for the eradication of H. pylori and it is significantly more effective in patients harbouring clarithromycin resistant strains.

The incidence side effects did not differ between therapy groups.

ELIGIBILITY:
Inclusion Criteria:

* Helicobacter pylori infected patients > 18 years

Exclusion Criteria:

* previous H. pylori eradication treatment;
* Use of proton pump inhibitors, H2-receptor antagonists, bismuth preparations and antibiotics in the previous 4 weeks;
* Concomitant anticoagulant or ketoconazole use, due to the potential of interaction with the study medications;
* Zollinger-Ellison syndrome;
* Previous surgery of the esophagus and/or upper gastrointestinal tract (with the exception of appendectomy, polypectomy and cholecystectomy);
* Severe or unstable cardiovascular, pulmonary, or endocrine disease; clinically significant renal or hepatic disease or dysfunction; hematological disorder; any other clinically significant medical condition that could increase the risk to the study participants; malignant disease of any kind during the previous 5 years except for successfully treated skin (basal or squamous cell) cancer or Barrett esophagus with high grade dysplasia;
* Drug or medication abuse within the past year;
* Severe psychiatric or neurological disorders;
* Pregnant or nursing women sexually active women of child bearing potential who were not willing to practice medically acceptable contraception (oral contraceptives; inject able/implantable or mechanical devices as well as vasectomy of the sexual partner) for the entire duration of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2003-07; Study Completion 2006-02

PRIMARY OUTCOMES:
13C urea breath test, upper endoscopy, histology, rapid urease test assessment

SECONDARY OUTCOMES:
bacterial culture, and antibiotic resistance assessment

CONTACTS AND LOCATIONS:
Overall Officials: Dino Vaira, M.D., Principal Investigator — S.Orsola/Malpighi Teaching Hospital, University of Bologna, Italy
Locations (1):
- S.Orsola/Malpighi Teaching Hospital, University, Bologna, Italy

REFERENCES:
- [Background] Zullo A, Gatta L, De Francesco V, Hassan C, Ricci C, Bernabucci V, Cavina M, Ierardi E, Morini S, Vaira D. High rate of Helicobacter pylori eradication with sequential therapy in elderly patients with peptic ulcer: a prospective controlled study. Aliment Pharmacol Ther. 2005 Jun 15;21(12):1419-24. doi: 10.1111/j.1365-2036.2005.02519.x. PMID 15948808
- [Background] De Francesco V, Margiotta M, Zullo A, Hassan C, Troiani L, Burattini O, Stella F, Di Leo A, Russo F, Marangi S, Monno R, Stoppino V, Morini S, Panella C, Ierardi E. Clarithromycin-resistant genotypes and eradication of Helicobacter pylori. Ann Intern Med. 2006 Jan 17;144(2):94-100. doi: 10.7326/0003-4819-144-2-200601170-00006. PMID 16418408
- [Derived] Vaira D, Zullo A, Vakil N, Gatta L, Ricci C, Perna F, Hassan C, Bernabucci V, Tampieri A, Morini S. Sequential therapy versus standard triple-drug therapy for Helicobacter pylori eradication: a randomized trial. Ann Intern Med. 2007 Apr 17;146(8):556-63. doi: 10.7326/0003-4819-146-8-200704170-00006. PMID 17438314